CLINICAL TRIAL: NCT04779528
Title: Awake Nasal Fiber-optic Intubation of Severely Obese Patients in Lateral Position: a Prospective Randomized Controlled Trial
Brief Title: Awake Nasal Fiber-optic Intubation of Severely Obese Patients in Lateral Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, omar ahmad ababneh, Principal investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 442/2021/67
Record Dates: First submitted 2021-02-27; First posted 2021-03-03 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Anesthesia; Intubation;Difficult; Intubation; Difficult or Failed; Anesthesia Intubation Complication
Keywords: Anesthesia; Intubation; obesity; fiberoptic
MeSH Terms: conditions — Obesity | interventions — Supine Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Patients will undergo fiberoptic intubation in supine position.
  Interventions: Procedure: Fiberoptic intubation in supine position.
- Group L (Experimental): Patients will undergo fiberoptic intubation in lateral position.
  Interventions: Procedure: Fiberoptic intubation in lateral position.

INTERVENTIONS:
Procedure: Fiberoptic intubation in supine position. — Patients will be placed in supine position after the establishment of full vital signs monitoring and the insertion of an intravenous line.
  Under sedation via intravenous infusion of remifentanil plus topical anesthesia with 10 ml of Lidocaine 1% via a 3.7mm bronchoscope. After applying a standard monitoring and preparation of the nose by decongestant and local anesthesia. A loaded flexible scope (by an endotracheal tube ETT) will be introduced through the nostril to reach the carina, then the ETT will be pushed over the scope 3cm above the carina.
  Arms: Group S
Procedure: Fiberoptic intubation in lateral position. — Patients will be placed in lateral position after the establishment of full vital signs monitoring and the insertion of an intravenous line.
  Under sedation via intravenous infusion of remifentanil plus topical anesthesia with 10 ml of Lidocaine 1% via a 3.7mm bronchoscope. After applying a standard monitoring and preparation of the nose by decongestant and local anesthesia. A loaded flexible scope (by an endotracheal tube ETT) will be introduced through the nostril to reach the carina, then the ETT will be pushed over the scope 3cm above the carina.
  Arms: Group L

SUMMARY:
Airway management in severely obese patients remains a challenging issue for anesthetists and may lead to life-threatening situations. Awake Fiber-Optic Bronchoscopy Intubation (FOBI) technique is considered as the gold standard when a difficult airway is anticipated to secure the airway and to facilitate the surgery. FOBI is usually done in supine position, while (in conscious patients) lateral position is the most recommended position to keep the upper airway patent. This prospective clinical trial study will test whether awake FOBI in Lateral position will provide a safe profile or a significant advantage over FOBI in supine position, in morbidly obese patients undergoing elective bariatric surgery.

DETAILED DESCRIPTION:
Airway management in severely obese patients remains a challenging issue for anesthetists and may lead to life-threatening situations. Awake Fiber-Optic Bronchoscopy Intubation (FOBI) technique is considered as the gold standard when a difficult airway is anticipated to secure the airway and to facilitate the surgery. FOBI is usually done in supine position, while (in conscious patients) lateral position is the most recommended position to keep the upper airway patent.

This prospective clinical trial study will test whether awake FOBI in Lateral position will provide a safe profile or a significant advantage over FOBI in supine position, in morbidly obese patients undergoing elective bariatric surgery. The main outcome is success rate and duration of the procedure. Secondary outcomes are oxygenation maintenance, hemodynamic stability, airway complication, sedation score, and postoperative airway morbidity in 6 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status classification two and three.
* Patients scheduled for elective bariatric surgeries under general anesthesia.

Exclusion Criteria:

* Refusal of fiberoptic intubation.
* Allergy to local anesthetics.
* Coagulopathy.
* Raised intracranial or intraocular pressure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
Duration of fiberoptic intubation. | 5 minutes
  The investigators will compare between the supine and lateral positions in terms of the duration needed for the insertion of an endotracheal tube via fiberoptic intubation.

SECONDARY OUTCOMES:
Complications during airway manipulation. | 5 minutes
  The investigators will document the occurrence of adverse events during fiberoptic intubation, and compare these complications between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No